CLINICAL TRIAL: NCT02887716
Title: Mapping the Lumbar Spine Marrow Adiposity
Acronym: FATFRAC
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: FATFRAC
Record Dates: First submitted 2016-08-30; First posted 2016-09-02 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Marrow Adiposity Lumbar Spine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to describe the change in the percentage of fat in the lumbar spine.

DETAILED DESCRIPTION:
The study of the distribution of bone marrow adiposity is little known in subjects who did not have pathology likely to alter the fat content of the vertebrae. Or that fat content is potentially a reflection of brittle bones (osteoporosis, for example), and deserves to be known because it can be used to normalize the lipid fraction values with respect to age or from the level (L1 , L2, L3, L4 or L5) of the vertebra being studied.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients who underwent MRI of the lumbar spine with Sagittal sequenceT1, T2 STIR and IDEAL, good quality, in a clinical setting type back pain, spondylitis research, radicular syndrome ...
* Examinations conducted between 2014 and 2015 on the same equipment
* Major patient
* Having formulated their non-opposition

Exclusion Criteria:

* Previous history of neoplastic disease
* Vertebral Fracture
* Pathology reaching the vertebral body detectable by MRI (disc lesion with rearrangements of the endplates (MODIC)
* Inflammation,
* Bone tumor,
* fracture
* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had an MRI of the lumbar spine in a context that justified (back pain, spondylitis research, radicular syndrome) having no corporeal spinal lesion at MRI examination.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Value of the fat fraction by vertebral level of the lumbar spine, in MRI, measured on the mapping generated by the IDEAL-IQ sequence. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Douraied Ben Salem, Professor, Principal Investigator — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France